CLINICAL TRIAL: NCT03433794
Title: Alcohol Health Education
Brief Title: Alcohol Health Education Among College Drinkers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abby Braitman (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Abby Braitman, Research Assistant Professor, Old Dominion University
Organization: Old Dominion University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-194; F32AA021310 (NIH)
Record Dates: First submitted 2018-02-08; First posted 2018-02-15 (Actual); Results first posted 2020-08-10 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: College Student Drinking
MeSH Terms: conditions — Alcohol Drinking in College | interventions — Ethanol; Immunization, Secondary

STUDY DESIGN:
Who Masked: Participant
Masking Description: The intervention is an online program, not an individual, so masking is not necessary. Similarly, the same online survey is deployed in all follow-up assessments regardless of condition, and data are not collected by individuals, so making is not necessary.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Placebo Comparator): The control group spent 60 minutes on an online education session (Lilly for Better Health) directed at other health behaviors besides alcohol. The site provides practical tips on general well-being such as healthy eating, physical activity, and stress management, as well as provides information on managing health conditions such as diabetes, heart disease and depression. Their email 2 weeks later contained only a reminder to participate in follow-up surveys.
  Interventions: Behavioral: Lilly for Better Health
- Intervention Only (Active Comparator): Participants navigated through Alcohol 101 Plus (TM) for 60 minutes. This is an online intervention, free to institutions and individuals. It is a combination of several intervention components, including alcohol education, personalized feedback, attitude-focused strategies, and skills training. It also included a virtual bar, where participants provide basic information such as sex, weight, and state of residence so that the program can provide tailored information on blood alcohol content (BAC) as well as state regulations regarding legal limits. Their email 2 weeks later contained only a reminder to participate in follow-up surveys.
  Interventions: Behavioral: Alcohol 101 Plus (TM)
- Intervention-plus-Booster (Experimental): Participants navigated through Alcohol 101 Plus (TM) for 60 minutes. This is an online intervention, free to institutions and individuals. It is a combination of several intervention components, including alcohol education, personalized feedback, attitude-focused strategies, and skills training. It also included a virtual bar, where participants provide basic information such as sex, weight, and state of residence so that the program can provide tailored information on blood alcohol content (BAC) as well as state regulations regarding legal limits. Importantly, their email 2 weeks later contained a reminder to participate in follow-up surveys, plus personalized feedback based on participant reported perceived alcohol norms, actual alcohol norms, and reported harm reduction strategies.
  Interventions: Behavioral: Alcohol 101 Plus (TM); Behavioral: Booster

INTERVENTIONS:
Behavioral: Alcohol 101 Plus (TM) — It is a combination of several intervention components, including alcohol education, personalized feedback, attitude-focused strategies, and skills training. It also included a virtual bar, where participants provide information such as sex, weight, and state so that the program can provide tailored information on blood alcohol content (BAC) as well as state regulations regarding legal limits. The program provides updated BACs based upon choices about what to consume and how quickly to consume it. The intervention is highly interactive, with text, photos, videos, and narratives for fictional students with decision points where the participant chooses what the fictional student should do. It is a non-linear environment, where participants choose which sections of the website to explore.
  Arms: Intervention Only; Intervention-plus-Booster
Behavioral: Booster — Personalized feedback was emailed to participants. Content included sex-specific descriptive normative information (i.e., drinks per week typically consumed by males and females at the same institution), as well as reminders of harm reduction strategies (i.e., techniques the participant reported using in their last survey, versus techniques not used).
  Other Names: Personalized Normative Feedback
  Arms: Intervention-plus-Booster
Behavioral: Lilly for Better Health — This is an online education session directed at other health behaviors besides alcohol. The site provides practical tips on general well-being such as healthy eating, physical activity, and stress management, as well as provides information on managing health conditions such as diabetes, heart disease and depression. It was not expected to influence alcohol use.
  Arms: Control

SUMMARY:
Alcohol use among college students is both widespread and problematic. There are many negative consequences associated with frequent alcohol use, ranging from mild (e.g., hangovers, missed classes) to severe (e.g., assault, even death). Online interventions targeting alcohol use among college students reduce alcohol consumption and associated problems. These interventions are popular among colleges because they are relatively inexpensive and easily disseminated. However, online interventions are not as efficacious as face-to-face interventions, such as brief motivational interviews. The proposed project employs emailed boosters in a randomized, controlled trial in an effort to improve the efficacy an existing, popular, free online intervention, while at the same time maintaining low cost and easy dissemination.

Adding boosters after interventions is a common technique to improve the efficacy of the original intervention. Boosters have been used successfully for alcohol use interventions among those seeking injury treatment in emergency medical settings. However, prior research has not supported booster efficacy for college student alcohol interventions. The current project develops and evaluates the effectiveness of boosters for a widely-used college student alcohol intervention. Specifically, the present project improves boosters by providing easy access via email; providing succinct, personalized feedback; and providing reminders of protective behavioral strategies. To test the effectiveness of adding boosters, participants randomized to alcohol-intervention-plus-boosters receive emails 2 weeks after the intervention with tailored feedback based upon their reported alcohol consumption. Participants are assessed up to nine months. The current research addresses the following specific aims:

Aim 1: Improve the efficacy of an easily-disseminated computerized intervention by adding personalized follow-up boosters, where efficacy is evidenced by reduced drinking and negative alcohol-related consequences (i.e., stronger effect sizes in the booster group immediately after receiving the booster).

Aim 2: Extend the duration of the reduction in drinking and associated problems through the use of these personalized follow-up boosters (i.e., significant differences between the booster and control groups at later timepoints).

Aim 3: Examine protective behavioral strategies highlighted by the booster as mediating behavioral mechanisms of change.

DETAILED DESCRIPTION:
Alcohol use within the college student population is both widespread and problematic. There are many negative consequences associated with frequent alcohol use, ranging from mild (e.g., hangovers, missed classes) to severe (e.g., assault, even death). College student alcohol use is a significant problem, and reducing consumption and associated problems is a priority among researchers, educators, and mental health professionals who work with this population.

Online interventions targeting alcohol use among college students reduce alcohol consumption and associated problems. These interventions are popular among colleges because they are relatively inexpensive and easily disseminated. However, online interventions are not as efficacious as face-to-face interventions, such as brief motivational interviews. The current project employs emailed boosters in a randomized, controlled trial in an effort to improve the efficacy an existing, popular, free online intervention, Alcohol 101 Plus (TM), while at the same time maintaining low cost and easy dissemination.

Adding boosters after interventions is a common technique to improve the efficacy of the original intervention. Boosters have improved the efficacy or effect duration for interventions targeting smoking cessation, mammograms, dating violence, caregiver skills, binge eating, and many other behaviors. Boosters have been used successfully for alcohol use interventions among those seeking injury treatment in emergency medical settings. Despite these successes, prior research has not supported booster efficacy for college student alcohol interventions. The current project develops and evaluates the effectiveness of boosters for a widely-used college student alcohol intervention by improving on the design of boosters. Specifically, the present project improves boosters by providing easy access via email to minimize burden; providing succinct, personalized feedback; and providing reminders of protective behavioral strategies. To test the effectiveness of adding boosters, participants randomized to the alcohol-intervention-plus-boosters condition receive emails 2 weeks after the intervention with tailored feedback based upon their reported alcohol consumption. Participants are initially assessed biweekly, then every three months up to nine months. The current research addresses the following specific aims:

Aim 1: Improve the efficacy of an easily-disseminated computerized intervention by adding personalized follow-up boosters, where efficacy is evidenced by reduced drinking and negative alcohol-related consequences (i.e., stronger effect sizes in the booster group immediately after receiving the booster).

Aim 2: Extend the duration of the reduction in drinking and associated problems through the use of these personalized follow-up boosters (i.e., significant differences between the booster and control groups at later timepoints after the significant differences between the intervention-only and control groups erode).

Aim 3: Examine protective behavioral strategies highlighted by the booster as mediating behavioral mechanisms of change.

3A: Determine if increased exposure to protective strategies through an emailed booster results in increased use of these strategies.

3B: Determine if those who increase their use of protective behavioral strategies decrease their alcohol consumption and related problems they experience.

3C: Assess the combination of these two effects (i.e., the indirect effect). The proposed study will be a critical first step to adapt existing online interventions. The findings from this study will be used to identify implications for modifying the protocol or booster.

ELIGIBILITY:
Inclusion Criteria:

* Current college students at the sponsor institution at the time of enrollment
* Between the ages of 18 and 24
* Consumed at least standard drink of alcohol in the past 2 weeks

Exclusion Criteria:

* Under age of 18
* Over age of 24
* Not a college student
* Did not drink alcohol in the past 2 weeks

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 537 (Actual)
Dates: Start 2013-01-29 (Actual); Primary Completion 2014-09-10 (Actual); Study Completion 2014-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abby L Braitman, Ph.D., Principal Investigator — Old Dominion University

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants read study description and eligibility criteria, and signed up to attend a baseline session. Upon joining the study and completing an informed consent document, they were randomly assigned to arm/group of the study. After completing the online survey, 26 individuals were identified as ineligible and not enrolled.
Groups:
- Intervention Only: Participants navigated through Alcohol 101 Plus (TM) for 60 minutes. Their email 2 weeks later contained only a reminder to participate in follow-up surveys.
  Alcohol 101 Plus (TM): It is a combination of several intervention components, including alcohol education, personalized feedback, attitude-focused strategies, and skills training. It also included a virtual bar, where participants provide information such as sex, weight, and state so that the program can provide tailored information on blood alcohol content (BAC) as well as state regulations regarding legal limits. The program provides updated BACs based upon choices about what to consume and how quickly to consume it. The intervention is highly interactive, with text, photos, videos, and narratives for fictional students with decision points where the participant chooses what the fictional student should do. It is a non-linear environment, where participants choose which sections of the website to explore.
- Intervention-plus-Booster: Participants navigated through Alcohol 101 Plus (TM) for 60 minutes. Importantly, their email 2 weeks later contained a reminder to participate in follow-up surveys, plus personalized feedback based on participant reported perceived alcohol norms, actual alcohol norms, and reported harm reduction strategies.
  Alcohol 101 Plus (TM): It is a combination of several components, including alcohol education, personalized feedback, attitude-focused strategies, and skills training. It also included a virtual bar, where the program can provide tailored information on blood alcohol content (BAC) as well as state regulations regarding legal limits. The intervention is highly interactive, with text, photos, videos, and narratives for fictional students with decision points where the participant chooses what the fictional student should do.
  Booster: Content included sex-specific descriptive normative information, as well as reminders of harm reduction strategies.
Period: Baseline
Arm/Group | Control | Intervention Only | Intervention-plus-Booster
Started | 183 | 173 | 181
Completed | 183 | 173 | 181
Not Completed | 0 | 0 | 0
Period: 2-Week Assessment
Arm/Group | Control | Intervention Only | Intervention-plus-Booster
Started | 183 | 173 | 181
Completed | 117 | 112 | 109
Not Completed | 66 | 61 | 72
Period: 4-Week Assessment
Arm/Group | Control | Intervention Only | Intervention-plus-Booster
Started | 183 | 173 | 181
Completed | 98 | 95 | 91
Not Completed | 85 | 78 | 90
Period: 6-Week Assessment
Arm/Group | Control | Intervention Only | Intervention-plus-Booster
Started | 183 | 173 | 181
Completed | 94 | 85 | 80
Not Completed | 89 | 88 | 101
Period: 3-Month Assessment
Arm/Group | Control | Intervention Only | Intervention-plus-Booster
Started | 183 | 173 | 181
Completed | 69 | 73 | 71
Not Completed | 114 | 100 | 110
Period: 6-Month Assessment
Arm/Group | Control | Intervention Only | Intervention-plus-Booster
Started | 183 | 173 | 181
Completed | 65 | 58 | 50
Not Completed | 118 | 115 | 131
Period: 9-Month Assessment
Arm/Group | Control | Intervention Only | Intervention-plus-Booster
Started | 183 | 173 | 181
Completed | 49 | 52 | 39
Not Completed | 134 | 121 | 142

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention Only | Intervention-plus-Booster | Total
Number analyzed (Participants) | 183 | 173 | 181 | 537
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.792 (1.779) | 19.792 (1.726) | 19.370 (1.476) | 19.650 (1.674)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 116 | 124 | 362
  Male | 61 | 57 | 57 | 175
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian or White | 82 | 92 | 88 | 262
  African-American or Black | 74 | 59 | 68 | 201
  Asian or Pacific Islander | 11 | 8 | 6 | 25
  Native American | 1 | 0 | 3 | 4
  Other | 10 | 10 | 14 | 34
  Hispanic | 24 | 18 | 13 | 55
  non-Hispanic | 158 | 154 | 167 | 479
Region of Enrollment [Number; unit: participants]
  United States | 183 | 173 | 181 | 537

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Consumption
Description: Participant self-reported number of standard drinks consumed by participant over the past 2 weeks
Time Frame: Past 2 weeks, reported at Baseline assessment (pre-intervention)
Measure: Mean (Standard Deviation); unit: drinks
Arm/Group | Control | Intervention Only | Intervention-plus-Booster
Number analyzed (Participants) | 183 | 173 | 181
drinks | 16.929 (14.826) | 17.988 (16.870) | 18.039 (16.382)

2. Secondary Outcome: Alcohol-related Consequences
Description: Participant self-report on the Young Adult Alcohol Consequences Questionnaire (YAACQ; Read, Kahler, Strong, & Colder, 2006), which assesses alcohol-related problems experienced by the participant. Total scores are created by summing all individual items, and range from 0 to 48, with higher values representing more problems experienced (i.e., worse outcomes).
Time Frame: Past 2 weeks, reported at Baseline assessment (pre-intervention)
Measure: Mean (Standard Deviation); unit: problems
Arm/Group | Control | Intervention Only | Intervention-plus-Booster
Number analyzed (Participants) | 183 | 173 | 181
problems | 6.656 (5.566) | 7.156 (6.066) | 7.011 (6.367)

ADVERSE EVENTS:
Arm/Group | Control | Intervention Only | Intervention-plus-Booster
All-Cause Mortality (participants affected / at risk) | 0/183 | 0/173 | 0/181
Serious Adverse Events (participants affected / at risk) | 0/183 | 0/173 | 0/181
Other Adverse Events (participants affected / at risk) | 0/183 | 0/173 | 0/181

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No